CLINICAL TRIAL: NCT01641783
Title: To Evaluate the Efficacy and Safety of ABI-007 Plus Capecitabine as First-line Chemotherapy for Advanced Gastric Cancer Patients:a Phase II Single Center Prospective Clinical Trial
Brief Title: Efficacy and Safety Study of ABI-007 Plus Capecitabine as First-line Chemotherapy for Advanced Gastric Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yanqiao Zhang (Other)
Responsible Party: Sponsor-Investigator, Yanqiao Zhang, Principal Investigator, The Third Affiliated Hospital of Harbin Medical University
Organization: The Third Affiliated Hospital of Harbin Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YL2012-03
Record Dates: First submitted 2012-07-11; First posted 2012-07-17 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Gastric Adenocarcinoma
Keywords: advanced; paclitaxel; capecitabine; first line therapy
MeSH Terms: interventions — Taxes; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- nanoparticle Albumin-bound paclitaxel (Experimental): evaluate one dose level of nab-paclitaxel:125mg/m2
  Interventions: Drug: nanoparticle Albumin-Bound paclitaxel

INTERVENTIONS:
Drug: nanoparticle Albumin-Bound paclitaxel — nanoparticle Albumin-Bound paclitaxel:125mg/m2 d1 iv
  Other Names: ABI-007

SUMMARY:
Gastric cancer remains one of the major causes of cancer deaths around the world,especially in Asia. For advanced gastric cancer,even if treated with chemotherapy,the prognosis is still poor, so the investigators urgently need an effective strategy to treat advanced gastric cancer, however, there was no recommended First-line chemotherapy for advanced gastric cancer. Taxane is promising in gastric cancer. Nanoparticle Albumin-Bound (Nab) Paclitaxel (Abraxane，ABI-007) with high effectiveness and low toxicity had been approved in breast cancer as first-line chemotherapy in many countries. The investigator then initiated a prospective phase II clinical trial with Nab-Paclitaxel plus Capecitabine as the first-line treatment in advanced gastric cancer to observe the efficacy and safety.

DETAILED DESCRIPTION:
A single arm,open,phase II study of Nab-Paclitaxel plus Capecitabine as the first-line treatment in advanced gastric cancer.

Nab-Paclitaxel should be given intravenously on days 1 and 8 at a dose as follows. Treatment should be repeated every 3 weeks:Nab-Paclitaxel:125 mg/m2; Capecitabine should be given orally twice a day as follows for 14 consecutive days, followed by a 1-week rest. Treatment should be repeated every 3 weeks. Capecitabine:1000mg/m2,twice daily (bid).

If applicable,the value of response and prognosis predictive factors are expected to be identified.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent form;
* histologically or cytologically confirmed gastric cancer;
* Age 18-75 years;
* Advanced or recurrent, metastatic disease;
* Performance Status- Eastern Cooperative Oncology Group (ECOG) 0-2;
* Life expectancy of at least 12 weeks;
* At least have one measurable disease(according to RECIST, Response Evaluation Criteria in Solid Tumors );
* no prior history of chemotherapy or beyond 6 months after the end of systemic adjuvant treatment;
* Haematopoietic status:

  * Absolute neutrophil count > 1.5 x 109/L;
  * Platelet count > 90 x 109/L;
  * Hemoglobin at least 90g/l;
* Hepatic status:

  * Bilirubin ≤ 1.5 x upper limit of normal (ULN);
  * AST and ALT ≤ 2.5 times ULN(no liver metastasis), ≤ 5 times ULN (with liver metastasis);
  * ALP ≤ 2.5 times ULN(no liver metastasis), ≤5 times ULN(with liver or bone metastasis);
  * serum albumin ≥ 30g/L;
* Renal status:

  * Creatinine ≤ 1.5 times ULN or calculated creatinine clearance, using the Cockcroft-Gault formula, ≥ 40 mL/min;
* Able to swallow and retain oral medication;

Exclusion Criteria:

* peripheral neuropathy of grade 2 or greater;
* symptomatic brain metastasis;
* known history of uncontrolled or symptomatic angina;
* clinically significant arrhythmias, congestive heart failure, uncontrolled hypertension (≥ 180/110), unstable diabetes mellitus, dyspnea at rest, or chronic therapy with oxygen;
* dementia, altered mental status, or any psychiatric condition that would prevent the understanding or rendering of ICF;
* active or uncontrolled infection;
* pregnant or lactating women;
* dysmetabolism with nanoparticle Albumin-bound paclitaxel or Capecitabine
* unable to swallow and retain oral medication,intestinal Obstruction,alimentary tract hemorrhage

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 1 year
  the follow-up visit of PFS will be performed every 6 weeks

SECONDARY OUTCOMES:
objective response rate | 6 weeks
  CT/MRI/Ultrasound will be performed every 2 cycles of treatment for efficacy evaluation
overall survival of participants | 2 years
  OS means that from the first dose of treatment drug to death or lost,the follow-up visit will be performed every 3 months till death or lost
biomarkers | 6 weeks
  To identify the molecular biomarkers(such as SPARK,β-Tubulin III,caveolin,etc)by immunohistochemical and western-bloting before and during therapy,to study the biomarkers correlations with clinical outcome and toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Yanqiao Zhang, M.D., Principal Investigator — Harbin Medical University